CLINICAL TRIAL: NCT06278857
Title: A Phase 2b, Open-label, Single Arm, Multicentre, Pilot Study of the Efficacy, Safety and Tolerability of Dostarlimab in Women With Early-stage MMR Deficient Endometrioid Endometrial Adenocarcinoma.
Brief Title: SATELLITE Study (feaSibility sAfeTy Efficacy dostarLimab earLy-stage defIcient endomeTrial cancEr)
Acronym: SATELLITE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Queensland Centre for Gynaecological Cancer (Other Government)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QCGC-001/2023
Record Dates: First submitted 2024-01-18; First posted 2024-02-26 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Endometrial Cancer Stage I; Mmr Deficiency; Endometrioid Endometrial Adenocarcinoma; Immune-related Adverse Event
Keywords: Endometrial Cancer Stage I; Mmr Deficiency; Immunotherapy drug; Anti-programmed death receptor - 1(PD-1)
MeSH Terms: conditions — Endometrial Neoplasms; Turcot syndrome | interventions — dostarlimab

STUDY DESIGN:
Intervention Model Description: This is a non-randomised, prospective, pilot, open-label, single arm study. Participation in this trial involves seven dostarlimab sessions over 12 months, with a treatment protocol of four cycles every three weeks, followed by a three-week break, and then three cycles every six weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single Arm (Experimental): Participation involves seven dostarlimab sessions over 12 months, with a treatment protocol of four cycles every three weeks, followed by a three-week break, and then three cycles every six weeks.
  Interventions: Drug: Dostarlimab-Gxly 50 MG/1 ML Intravenous Solution [JEMPERLI]

INTERVENTIONS:
Drug: Dostarlimab-Gxly 50 MG/1 ML Intravenous Solution [JEMPERLI] — The dosing regimen follows standard clinical care protocol comprising of 4 cycles every 3-weeks, a rest period of 34 weeks followed by 3 cycles every 6 weekly for a total of 7 cycles.
  Other Names: JEMPERLI

SUMMARY:
The main goal of this clinical trial is to evaluate dostarlimab, an immunotherapy drug, as a potential alternative to surgery for early-stage endometrial cancer with Mismatch Repair deficiency, a genetic cause for 20-30% of cases. The study aims to establish dostarlimab's efficacy and safety in early-stage endometrial cancer, exploring its potential as a non surgical option for those unsuitable or unwilling to undergo major surgery, allowing for fertility preservation or addressing specific health conditions.

Participants will have seven dostarlimab sessions over 12 months. The treatment plan involves four cycles every three weeks, followed by a three-week break, and then three cycles every six weeks.

This research is a promising step toward a new, less invasive treatment choice for patients with specific genetic traits. It expands the range of care options for endometrial cancer.

DETAILED DESCRIPTION:
Cancer of the endometrium is a common type of cancer that affects over 3,000 women in Australia every year. The usual way to treat this cancer is by having surgery to remove the uterus, fallopian tubes, ovaries, and sometimes lymph nodes. But this surgery might not be the best choice for women who want to have children or for older women, those with obesity, or people with other health problems, because surgery can be risky for them.

Big improvements in the treatment of endometrial cancer have occurred due to new technology and enhanced understanding of this cancer. In the past, doctors decided how to treat this cancer based on what it looked like and how likely it was to come back. But in recent years, they've been looking at the genes of the cancer to figure out the best treatment for each person. This is important to make sure each patient gets the right care.

The research project evaluates dostarlimab, an immunotherapy drug, as a potential alternative to surgery for early-stage endometrial cancer with Mismatch Repair deficiency, a genetic cause for 20-30% of cases. DNA repair errors can lead to cancer, and the Mismatch Repair (MMR) pathway addresses these errors. dostarlimab enhances the immune system's ability to combat cancer by blocking specific proteins, and while approved in Australia for advanced cases, its effectiveness in early-stage cancer is unknown. The study aims to establish dostarlimab's efficacy and safety in early-stage endometrial cancer, exploring its potential as a non-surgical option for those unsuitable or unwilling to undergo major surgery, allowing for fertility preservation or addressing specific health conditions. The study proposes a unique approach to endometrial cancer treatment.

Participation involves seven dostarlimab sessions over 12 months, with a treatment protocol of four cycles every three weeks, followed by a three-week break, and then three cycles every six weeks.

Dostarlimab is approved in Australia for the treatment of adult patients with recurrent or advanced mismatch repair deficient endometrial cancer. However, it is not currently approved to treat early-stage endometrial cancer. This study will test to see if dostarlimab is an effective treatment for early-stage mismatch repair deficient endometrial cancer. Dostarlimab may be a good option for women who cannot or do not want to have surgery to remove their uterus, fallopian tubes, ovaries and lymph nodes, or who want to keep the option of having children.

This research offers hope for a novel, non-invasive treatment option for patients with specific genetic characteristics, expanding the scope of endometrial cancer care.

Primary objective: To determine the absence of endometrial cancer following protocol treatment regimen of dostarlimab

Secondary objective: To determine the safety and tolerability of dostarlimab in participants with early-stage MMR deficient endometrioid endometrial adenocarcinoma

Exploratory Objective:

* To assess study feasibility
* Assess participant evaluation of study participation providing consumer feedback to inform future clinical research programs.
* To assess longer term (9 and 12 months) changes to laboratory and clinical parameters post treatment with dostarlimab.
* Exploratory investigations utilizing biobanked tissue, blood samples for participant treated with dostarlimab.
* An exploratory outcome of increased clinical efficacy (pCR) related to irAEs.
* Fertility Outcome

ELIGIBILITY:
Inclusion Criteria:

1. Female participant is at least 18 years of age (at the time of informed consent).
2. Participant has:

   i. histologically or cytologically proven Stage 1, FIGO grade 1 or 2, MMR deficient (Absence of at least one MMR protein (MLH1, PMS2, MSH2, MSH6) by immunohistochemistry.) endometrioid endometrial adenocarcinoma, and

   ii. wish to preserve the uterus or are not a suitable candidate for hysterectomy.
3. Participant has an ECOG performance status of ≤ 2
4. Participant demonstrates no evidence of extrauterine disease assessed from all available clinical evidence (physical examination findings) and medical imaging including standard of care diagnostic CT, MRI, ultrasound, or X-ray and screening gadolinium contrast pelvic MRI
5. Participants must have adequate organ and bone marrow function defined as:

   i. absolute neutrophil count 1.5 x 109/L ii. platelets 100 x 109/L iii. haemoglobin ≥9 g/dL

   Adequate liver function:

   iv. total bilirubin < 1.5x institutional upper limit normal (ULN) v. AST/ALT < 2. 5 - 3x ULN

   Adequate renal function as defined by:

   vi. Creatinine < 1.5x institutional upper limits OR creatinine clearance > 30 ml/min

   Adequate coagulation profile:

   vii. INR or PT ≤ 1.5 x ULN unless the participant is receiving anticoagulant therapy as long as INR or PTT is within the therapeutic range of intended use of anticoagulants viii. aPTT ≤ 1.5 x ULN unless the patient is receiving anticoagulant therapy as long as INR or PTT is within the therapeutic range of intended use of anticoagulant
6. A potential participant with a clinical abnormality or laboratory parameters outside the normal reference range for the population being studied may be rescreened once, at the Investigator's discretion, and may be included only if the Investigator considers that the finding is unlikely to introduce additional risk factors to the participant and will not interfere with the study procedures.
7. Women of child-bearing potential (WOCBP) must have a negative serum pregnancy test at enrolment prior to each treatment cycle and use a highly effective contraceptive method including; oral contraceptive pills [OCPs], or an intrauterine hormone device [IUD]) from screening until at least 4 months following the last dose of dostarlimab. Females who are abstinent from heterosexual intercourse as part of their usual lifestyle do not need to use contraception.
8. Post-menopausal females. Post-menopausal status will be confirmed through testing of follicle-stimulating hormone (FSH) levels (≥ 40 IU/mL) at screening for amenorrhoeic (≥ 12 months) female participants.
9. Participants with confirmed Type I or Type II diabetes mellitus must be well controlled by medication and/or diet and have glycated haemoglobin (HBAc1) < 8.5% at screening and be willing to monitor blood glucose levels at home during study participation.
10. Participants must have normal blood pressure (BP) or adequately treated and controlled hypertension.
11. Participant is able to provide written informed consent and are willing to participate for the duration of the study and to follow study procedures.

Exclusion Criteria:

1. Participant has a histological (cell) type other than endometrioid adenocarcinoma (sarcomas or high-risk endometrial e.g., papillary serous, clear cell).
2. Participant is pregnant, breastfeeding, or planning to become pregnant during the trial period.
3. Participant has had an allogeneic tissue/solid organ transplant.
4. Participants with uncontrolled hypertension, history of hypertension crisis, history of hypertensive encephalopathy, QTc>450 at baseline, other severe cardiovascular diseases including cerebrovascular accident (CVA), transient ischemic attack (TIA), myocardial infarction (MI), unstable angina, New York Heart Association (NYHA) class III and IV heart failure and uncontrolled arrhythmia within the past 6 months. Rate-controlled arrhythmia may be eligible at the discretion of the Investigator.
5. Participant is considered a poor medical risk due to an uncontrolled medical disorder, non-malignant systemic disease, or active infection (including, r acute pelvic inflammatory disease), requiring intravenous antibiotics within the past 2 weeks. Specific examples include, but are not limited to, active, non-infectious pneumonitis; uncontrolled major seizure disorder; unstable spinal cord compression; superior vena cava syndrome; or any psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study (including obtaining informed consent).
6. Participant has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days before the study start.
7. Participant has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with the use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Use of inhaled steroids, local injection of steroids, and steroid eye drops are allowed.
8. Participant with severe acute respiratory syndrome coronavirus 2 (SARS- CoV-2; COVID-19) influenza A/B within 3 months of screening.
9. Participant received a transfusion of blood products (including platelets or red blood cells) within 21 days prior to the first dose of the study drug.
10. Participant has undergone major surgery in the 4 weeks prior to consent.
11. Participant has -experienced any of the following with prior immunotherapy: any immune-related AE (irAE) of Grade 3 or higher, immune-related severe neurologic events of any grade (e.g., myasthenic syndrome/myasthenia gravis, encephalitis, Guillain-Barré Syndrome, or transverse myelitis), exfoliative dermatitis of any grade (Stevens-Johnson Syndrome, toxic epidermal necrolysis, or drug reaction with eosinophilia and systemic symptoms [DRESS] syndrome), or myocarditis of any grade. Non-clinically significant laboratory abnormalities are not exclusionary.)
12. Participant has taken part in a clinical trial of an investigational medical product or device within 30 days or 5 half-lives before study start, whichever comes later. [except hormonal IUD]
13. Participant has a concomitant malignancy, or participant has a prior non-endometrial invasive malignancy who has been disease-free for ≤5 years since end of treatment for the malignancy Non-melanoma skin cancer and definitively treated in-situ carcinomas is allowed.
14. Participant has a known history of Human Immunodeficiency Virus (HIV), or a positive test at screening.
15. Known active Hepatitis B or C, complete curative treatment and have no detectable viral RNA.
16. Participants are known to be hypersensitive to the active substance or any of the excipients.
17. Participant has a history or current diagnosis of interstitial lung disease.
18. Participant has received or is scheduled to receive, a live vaccine within 30 days before the first dose of study treatment, during study treatment, and for up to 180 days after receiving the last dose of study treatment.
19. Unwilling or unable to follow protocol requirements, including attendance at follow-up visit/s.
20. Participant has any condition contraindicated with tumor /blood sampling procedures required by the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Determine the absence endometrial cancer following protocol treatment regimen of dostarlimab. | Week 27 (Month 6)
  Number of participants achieving investigator-assessed pathological complete response (pCR).

SECONDARY OUTCOMES:
Determine the safety and tolerability of dostarlimab in participants with early-stage MMR deficient endometrioid endometrial adenocarcinoma. | From Cycle 1 /Day 1 to 30 days post last dose, 9 and 12months.
  Safety analyses including incidence of treatment-emergent adverse events (TEAEs), immune-related AEs of interest (irAEIs), and serious adverse events (SAEs), toxicities graded 3-5 as per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version 5.0).
TEAEs/irAEIs Leading to Study Drug Discontinuation | Screening to Cycle 7 (Week 25)
  Explore the frequency and severity of TEAEs/irAEIs that lead to discontinuation of the study drug.
TEAEs/irAEIs Leading to Study Withdrawal | From Screening to Week 27 (6 months) 9 and 12months.
  Investigate and assess the frequency and severity of TEAEs/irAEIs resulting in the withdrawal of participants from the study.
Clinically Significant Changes in Haematology | From Screening to Week 27 (6 months) 9 and 12months to End of Study.
  Assess the number of participants with clinically significant changes in Haematology
Clinically Significant Changes in Clinical Chemistry | From Screening to Week 27 (6 months) 9 and 12months to End of Study.
  Assess the number of participants with clinically significant changes in Clinical Chemistry
Clinically Significant Changes in Thyroid Function | From Screening to Week 27 (6 months)
  Assess the number of participants with clinically significant changes in Thyroid Function (Measure thyroid-stimulating hormone (TSH), free thyroxine (FT4), and triiodothyronine (T3) levels.)
Abnormal Vital Signs | From Screening to Week 27 (6 months) 9 and 12months.
  Assess the number of participants with abnormal vital signs pre and post treatment.
Abnormal Electrocardiogram (ECG) Parameters | Screening, Week 12 (3 months) and Week 27 (6 months)
  Asses the number of participants with abnormal ECG parameters.
Clinically Significant Abnormal Physical Examination | From screening visit to Week 27 (6 months), 9 and 12 months
  Assess the number of participants with clinically significant abnormal physical examinations.
Concomitant Medications | From Screening to 12 months.
  Assess the number of participants who are taking concomitant medications

OTHER OUTCOMES:
Study Feasibility Outcome: Recruitment Rate | 2 Years
  Evaluates the pace of participant recruitment in the study by comparing the number of enrolments per time unit with the set recruitment objectives.
Study Feasibility Outcome: Rationale for Treatment Discontinuation | through study completion, an average of 2 year
  Evaluates the number of participants who withdraw from the study and the reasons behind treatment discontinuation.
Study Feasibility Outcome: Study Withdrawal Rate | through study completion, an average of 2 year
  Calculate the percentage of participants who withdraw from the study, irrespective of the reason, to understand the overall attrition rate.
Study Feasibility Outcome: Incidence of Immune-Related Adverse Events (irAEs) | At the end of cycle 1 to 4 (each cycle is 21 days) and cycle 5 to 7 (each cycle is 42 days)
  Calculate the ratio of participants experiencing irAEs to the total number of participants, providing insights into the safety profile of the treatment.
Study Feasibility Outcome: Number of Cycles of dostarlimab Completed | through study completion, an average of 2 year
  Count the total number of treatment cycles completed by participants, indicating the adherence and completion rates of the dostarlimab regimen.
Qualitative Evaluation by Semi-Structured Interview to gather valuable consumer feedback to inform future clinical research programs. | 12 month
  Conducting semi-structured interviews with participants to gain insights into their perceptions, facilitators, and barriers related to study participation.
Participant Burden Assessment | 12 months
  Assess the perceived burden related to the clinical procedures and treatment protocols imposed on participants throughout the study by collecting feedback on the challenges and difficulties participants face in adhering to the clinical procedures and treatment protocols, quantifying the perceived burden.
Participant Burden Assessment - Adverse Events | 12 months
  Evaluate the impact of adverse events on participants' experiences and well-being during the course of the study by capturing participants' feedback on the severity and frequency of adverse events, providing a comprehensive understanding of the burden associated with these events.
Evaluation of Fertility Outcomes/Pregnancy Plans for WOCBP compare to their pre-treatment reproductive plans. | 12 months
  Compare the participants' pre-treatment reproductive plans with the actual fertility outcomes and pregnancy plans, providing insights into the impact of the study on these important aspects of participants' lives.
Correlate clinical efficacy (pCR) with irAEs. | Week12 (3 months), Week 27 (6 months) and 12 months.
  Time change course of pCR and irAEs.
Fertility outcome within the fertility preservation population - pregnancy rates | 24 months
  Evaluate pregnancy rates within the fertility preservation population.
Fertility outcome within the fertility preservation population - pregnancy loss rates | 24 months
  Evaluate pregnancy loss rates within the fertility preservation population.
Fertility outcome within the fertility preservation population - live birth rates | 24 months
  Evaluate live birth rates within the fertility preservation population.
Fertility outcome within the fertility preservation population - rates of maternal and fetal complications/abnormalities | 24 months
  Evaluate rates of maternal and fetal complications/abnormalities within the fertility preservation population.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Obermair, Professor, Study Chair — Queensland Centre for Gynaecological Cancer (QCGC) Research
Locations (3):
- Australia (3):
  - Westmead Hospital, Sydney, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Obermair A, Gebski V, Goh J, Kuchel A, Brand A, Mak B, McNally O, Baxter E, Jobling T, Mileshkin L. Phase 2b, open-label, single-arm, multicenter pilot study of the efficacy, safety, and tolerability of dostarlimab in women with early-stage mismatch repair-deficient endometrioid endometrial adenocarcinoma. Int J Gynecol Cancer. 2025 Apr;35(4):101644. doi: 10.1016/j.ijgc.2025.101644. Epub 2025 Jan 16. PMID 39955187